CLINICAL TRIAL: NCT05627362
Title: A Phase II, Multicenter, Double-Blind, Randomised, Placebo-Controlled Study and Open Label Long Term Extension to Evaluate the Safety and Efficacy of Elafibranor in Adult Participants With Primary Sclerosing Cholangitis (PSC).
Brief Title: A Study to Assess Safety and Effectiveness of Elafibranor in Adult Participants With Primary Sclerosing Cholangitis.
Acronym: ELMWOOD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-60190-453; 2022-002695-37 (EudraCT Number)
Record Dates: First submitted 2022-11-22; First posted 2022-11-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double-Blind Period: Elafibranor 80 mg (Experimental): Participant will receive two tablets per day (one tablet of elafibranor 80 mg + 1 tablet of placebo matching the 120 mg sized tablet) over the 12 weeks in Double-blind period.
  Interventions: Drug: Elafibranor 80 mg; Drug: Placebo Matched to Elafibranor 120 mg
- Double-Blind Period: Elafibranor 120 mg (Experimental): Participant will receive 2 tablets per day (one tablet of elafibranor 120 mg + 1 tablet of placebo matching the 80 mg sized tablet) over the 12 weeks in Double-blind period.
  Interventions: Drug: Elafibranor 120 mg; Drug: Placebo Matched to Elafibranor 80 mg
- Double-Blind Period: Placebo (Placebo Comparator): Participant will receive 2 placebo tablets per day (one matching the 80 mg sized tablet + one matching the 120 mg sized tablet) over the 12 weeks in Double-blind period.
  Interventions: Drug: Placebo Matched to Elafibranor 80 mg
- Open-Label Extension Period: Elafibranor 120 mg (Experimental): Participant will receive one tablet per day (elafibranor 120 mg) over the 96 weeks in Open-Label extension period.
  Interventions: Drug: Elafibranor 120 mg

INTERVENTIONS:
Drug: Elafibranor 80 mg — Oral Tablet
  Other Names: GFT505
  Arms: Double-Blind Period: Elafibranor 80 mg
Drug: Elafibranor 120 mg — Oral Tablet
  Other Names: GFT505
  Arms: Double-Blind Period: Elafibranor 120 mg; Open-Label Extension Period: Elafibranor 120 mg
Drug: Placebo Matched to Elafibranor 80 mg — Oral Tablet
  Arms: Double-Blind Period: Elafibranor 120 mg; Double-Blind Period: Placebo
Drug: Placebo Matched to Elafibranor 120 mg — Oral Tablet
  Arms: Double-Blind Period: Elafibranor 80 mg

SUMMARY:
This study will evaluate the effects of elafibranor (the study drug) in participants with Primary Sclerosing Cholangitis (PSC). PSC is a rare disease of the liver that leads to injury and destruction of bile ducts. Damage to bile ducts leads to buildup of bile in the liver, which then causes further damage, and leads to disease progression. This study will compare elafibranor to a placebo, a dummy treatment. The main objective of the trial will be to study the safety and side effects of the study drug. The trial will also study the study drug's effects on blood tests and other tests related to PSC disease activity.

ELIGIBILITY:
Inclusion Criteria :

* Participants with a diagnosis of Primary sclerosing cholangitis (PSC) as demonstrated by the presence of the following, and in the absence of apparent causes of secondary sclerosing cholangitis: i) Historical evidence of an elevated Alkaline phosphatase (ALP) > Upper Limit Normal (ULN) since at least 6 months prior to SV1. ii) Cholangiogram (e.g. magnetic resonance cholangiopancreatography (MRCP), endoscopic retrograde cholangiopancreatography (ERCP), percutaneous transhepatic cholangiography (PTC) with features compatible with large duct PSC.
* ALP ≥1.5x ULN during screening (with variability ≤30% based on two values).
* Total bilirubin ≤2.0x ULN at Screening Visit 1(SV1)
* Participants taking ursodeoxycholic acid (UDCA) at a total daily dose ≤23 mg/kg/day, with a minimum of 6 months of stable treatment prior to screening period and expected to remain on stable dose through the 12-week DBP. Minimum of 3 months off treatment prior to screening period if UDCA was recently discontinued.
* For participants with Inflammatory bowel disease (IBD): i) Participants with Crohn's disease must be in remission based on the investigator's clinical assessment and should be on stable treatment prior to randomisation and during screening. ii) Participants with ulcerative colitis must be in remission or have low activity disease as per the judgement of the investigator and should be on stable treatment prior to randomisation and during screening. iii) Current treatment for IBD is permitted, if the participant has been well controlled for ≥3 months prior to the screening period and is anticipated to remain on a stable dose of drugs for IBD treatment, including biologics, immunosuppressants, immunomodulators, or systemic corticosteroids. iv) Participants with IBD should have a colonoscopy performed within one year prior to the screening period showing no evidence of dysplasia or cancer.
* Medications for management of pruritus (e.g. cholestyramine, rifampin, naltrexone or sertraline) must be on a stable dose for ≥3 months prior to the screening period.
* Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. -A female participant is eligible to participate if she is not pregnant or breastfeeding at screening, is willing not to become pregnant during the study and is willing to follow applicable protocol requirements related to this. - Male participants are eligible to participate if they agree to follow applicable protocol requirements related to contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria :

* History or presence of other concomitant chronic liver disease including: i) ImmunoglobulinG 4 (IgG4) related sclerosing cholangitis, or IgG4 ≥4x ULN at SV1. ii) Small duct PSC. iii) Documented history of secondary sclerosing cholangitis. iv) Presence of hepatitis B surface antigen (HBsAg) at screening. v) Hepatitis C virus (HCV) infection vi) Primary biliary cholangitis (PBC) or positive anti-mitochondrial antibody. vii) Alcohol-related liver disease. viii) Autoimmune hepatitis (AIH): Simplified Diagnostic Criteria of the IAIHG ≥6. ix) Presence of history of PSC-PBC or PSC-AIH overlap syndrome. x) Non-alcoholic steatohepatitis (NASH). SMD form protocol master data--23- INT / Version 1 Known history of alpha-1 antitrypsin deficiency
* Presence of percutaneous drain or bile duct stent at screening or within three months prior to screening.
* History of bacterial cholangitis within 60 days prior to the screening period, or participant on antibiotics for prophylaxis of recurrent cholangitis.
* History or any current suspicion of cholangiocarcinoma or elevated value of carbohydrate antigen 19-9 (CA19-9) >129 U/mL at SV1.
* Alpha-fetoprotein (AFP) >20 ng/mL with 4-phase liver computerised tomography (CT) or magnetic resonance imaging (MRI) suggesting presence of liver cancer.
* Participants with cirrhosis who are also classified as Child-Pugh B or C based on the Child-Pugh score. Participants with cirrhosis with Child-Pugh A score are allowed.
* History of clinically significant hepatic decompensation as described in the study protocol
* Presence or history of hepatocellular carcinoma.
* Medical conditions that may cause non-hepatic increases in ALP (e.g. Paget's disease).
* Medical conditions that may diminish life expectancy to <2 years, including known cancers.
* Participant has a positive test for human immunodeficiency virus (HIV) type 1 or 2 at SV1, or participant is known to have tested positive for HIV.
* Evidence of any other unstable or untreated clinically significant immunological, endocrine, neurological, gastrointestinal, haematologic, psychiatric diseases as evaluated by the investigator; other clinically significant conditions that are not well controlled
* Known malignancy or history of malignancy within the last 5 years, with the exception of local, successfully treated basal cell carcinoma or in-situ carcinoma of the uterine cervix.
* Participants with previous exposure to elafibranor
* ALT and/or AST >5x ULN
* Albumin <3.0 g/dL at SV1.
* Platelet count <100,000/microliter.
* International normalised ratio (INR) >1.3 due to altered hepatic function.
* Creatine phosphokinase (CPK) >2x ULN during screening period.
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment Emergent Adverse Event (TEAEs), Treatment Related TEAEs, Serious Adverse (SAEs) and Adverse Events of Special Interest (AESIs) | Double Blind Period: Baseline up to week 12, Open Label Extension (OLE) Period: Baseline up to week 100
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AESIs are AEs that may not be serious but are of special importance to a particular drug or class of drugs.
Percentage of Participants With Clinically Significant Changes in Physical Examination Findings | Double Blind Period: Baseline up to week 12, OLE Period: Baseline up to week 100
  Percentage of participants with clinically significant changes in physical examination findings will be reported. The clinical significance will be decided by the investigator.
Percentage of Participants With Clinically Significant changes in Laboratory Parameters (blood chemistry, hematology and coagulation) | Double Blind Period: Baseline up to week 12, OLE Period: Baseline up to week 100
  Percentage of participants with clinically significant change in laboratory parameters (blood chemistry, hematology and coagulation) will be reported. The clinical significance will be decided by the investigator.
Percentage of Participants With Clinically Significant Changes in Vital Signs | Double Blind Period: Baseline up to week 12, OLE Period: Baseline up to week 100
  Percentage of participants with clinically significant changes in Vital Signs will be reported. The clinical significance will be decided by the investigator.
Percentage of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Readings | Double Blind Period: Baseline up to week 12, OLE Period: Baseline up to week 100
  Percentage of participants with clinically significant changes in ECG readings will be reported. The clinical significance will be decided by the investigator.

SECONDARY OUTCOMES:
Relative Change From Baseline in Alkaline Phosphate Levels (ALP) | Double Blind Period: Baseline, Week 12, OLE Period: Baseline, Week 52, Week 96
Percentage of Participants With ≥40% Decrease from Baseline in ALP Levels | Double Blind Period: Baseline, Week 12, OLE Period: Baseline, Week 52, Week 96
Absolute Change from Baseline in ALP | Double Blind Period: Baseline, Week 12, OLE Period: Baseline, Week 52, Week 96
Percentage of Participants With ALP: <1.3x Upper Limit of Normal (ULN) and <1.5x ULN | Double Blind Period: Week 12
Percentage of Participants who Normalised ALP | Double Blind Period: Week 12
Change From Baseline in Alanine Transaminase (ALT),Aspartate Transaminase (AST), Gamma-glutamyl transferase (GGT), 5' Nucleotidase and Fractionated ALP Levels at Week 12 | Baseline, Week 12
Change From Baseline in Total bilirubin, Conjugated bilirubin Levels at Week 12 | Baseline, Week 12
Change From Baseline in Albumin Levels at Week 12 | Baseline, Week 12
Change from Baseline in Enhanced Liver Fibrosis (ELF) Test Score | Double Blind Period: Baseline, Week 12
Change From Baseline in Liver Stiffness Measurement (LSM) Values Assessed by FibroScan® at Week 12 | Double Blind Period: Baseline, Week 12
Change From Baseline in Other Non-invasive Hepatic Fibrosis Serum Markers as Measured by PAI-1, TGF-β, Marker of type V Collagen Formation (Pro-C5), and Marker of Type III Collagen Formation (Pro-C3) | Double Blind Period: Baseline, Week 12
Change From Baseline in Fibrosis-4 (FIB-4) and AST to Platelet Ratio Index (APRI) | Double Blind Period: Baseline, Week 12
Change From Baseline in Cytokeratin-18 (CK-18) (M65 and M30) Levels | Double Blind Period: Baseline, Week 12
Pharmacokinetics (PK) of Elafibranor and its Metabolite GFT1007: Area Under the Concentration-time Curve Over the Dosing Interval from Time 0 to 24 hours(AUC0-24) | Pre-dose, 0.5 hour (h), 1h, between 1.5 hours and 2h, 4h, and 6h after dosing at Week 4
  AUC 0-24 will be recorded from the PK blood samples collected.
PK of Elafibranor and its Metabolite GFT1007: Maximum (peak) Observed Plasma Drug Concentration (Cmax) | Pre-dose, 0.5 hour (h), 1h, between 1.5h and 2h, 4h, and 6h after dosing at Week 4
PK of Elafibranor and its Metabolite GFT1007: Time to Maximum Observed Drug Concentration (Tmax) | Pre-dose, 0.5 hour (h), 1h, between 1.5h and 2h, 4h, and 6h after dosing at Week 4
  Tmax will be recorded from the PK blood samples collected.
PK of Elafibranor and its Metabolite GFT1007: Total Body Clearance (Cl/F) | Double Blind Period: Baseline up to Week 12
  Cl/F will be recorded from the PK blood samples collected.
PK of Elafibranor and its Metabolite GFT1007: Volume of distribution (Vz) | Double Blind Period: Baseline up to Week 12
  Vz will be recorded from the PK blood samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical, Director, Study Director — Ipsen
Locations (62):
- United States (30):
  - Om Research LLC, Lancaster, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - Sutter Health Van Ness Campus Medical Office Building, San Francisco, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - South Denver Gastroenterology,P.C., Englewood, Colorado
  - Rocky Mountain Gastroenterology (RMG), Littleton, Colorado
  - Yale University School Of Medicine - Yale Center For Clinical Investigation, New Haven, Connecticut
  - Schiff Center for Liver Diseases - University of Miami, Miami, Florida
  - Covenant Research, Sarasota, Florida
  - Piedmont Hospital - Piedmont Transplant Institute, Atlanta, Georgia
  - Tandem Clinical Research GI, Marrero, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Liver Research Center, Boston, Massachusetts
  - Huron Gastroenterology Associates - Center for Digestive Care, Ypsilanti, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Southwest Gastroenterology Associates, PC (SWGA), Albuquerque, New Mexico
  - New York University Langone Health, New York, New York
  - Gastro Health Research, Cincinnati, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Gastro One, Cordova, Tennessee
  - University Of Texas Southwestern Medical Center At Dallas, Dallas, Texas
  - American Research Corporation at The Texas Liver Institute, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Bon Secours Richmond Community Hospital LLC. d/b/a Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University Of Alberta Hospital-Zeidler Ledcor Centre, Edmonton, Alberta
  - Brampton Civic Hospital (BCH) - Osler Hepatitis Centre, Brampton, Ontario
  - Aspen Woods Clinic, Calgary
  - Centre de Recherche du Centre Hospitalier de l'Universite de Montreal, Montreal
  - G.I Research Institute, Vancouver
- Germany (4):
  - Charite Campus Virchow, Berlin
  - Klinikum der Johann Wolfgang Goethe-Universitaet Frankfurt, Frankfurt
  - Universitaetsklinikum Heidelberg - Nationales Centrum fuer Tumorerkrankungen, Heidelberg
  - University Hospital Ulm, Ulm
- Italy (5):
  - Azienda Ospedaliero Universitaria Modena, Modena
  - Azienda Ospedaliera di Padova - U.O.C. di Gastroenterologia, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Gruppo Humanitas - Humanitas Research Hospital, Istituto Clinico Humanitas, Rozzano
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Portugal (3):
  - Centro Hospitalar do Alto Ave - Hospital Senhora da Oliveira, Guimarães
  - Centro Hospitalar Universitario Lisboa Norte, Lisbon
  - Centro Hospitalar de Lisboa ocidental (CHLO), Hospital Egas Moniz, Lisbon
- Spain (7):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon (HGUGM), Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital De Montecelo, Pontevedra
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (7):
  - Aberdeen Royal Infirmary NHS Grampian Grampian Health Board, Aberdeen
  - Queen Elizabeth Hospital, Birmingham
  - Frimley Park Hospital - Frimley Health NHS Foundation Trust, Frimley
  - Glasgow Royal Infirmary - Greater Glasgow Health Board, Glasgow
  - Hull Royal Infirmary - Hull University Teaching Hospitals NHS Trust, Hull
  - Ambrose King Centre-Royal London Hospital-Barts Health NHS Trust, London
  - The Royal Free Hospital - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/

REFERENCES:
- [Derived] Levy C, Abouda GF, Bilir BM, Bonder A, Bowlus CL, Campos-Varela I, Cazzagon N, Chandok N, Cheent K, Cortez-Pinto H, Demir M, Dill MT, Eksteen B, Fenkel JM, Gilroy R, Ko HH, Jacobson IM, Kallis Y, Kugelmas M, Luketic V, Mangia A, Montano-Loza AJ, Mukhopadhya A, Olveira A, Patel BC, Pietrangelo A, Pradhan F, Salcedo M, Shiffman ML, Sprinzl K, Swann R, Thorburn D, Thuluvath PJ, Trivedi PJ, Turnes J, Zein CO, Gomes da Silva H, Jaitly S, Miller B, Milligan C, Tavenard A, Kowdley KV. Safety and efficacy of elafibranor in primary sclerosing cholangitis: The ELMWOOD phase II randomized-controlled trial. J Hepatol. 2026 Jan;84(1):74-85. doi: 10.1016/j.jhep.2025.04.025. Epub 2025 May 10. PMID 40350321